CLINICAL TRIAL: NCT02812602
Title: Topical Anesthesia With Lidocaine Patch for Removal of Metal Staples After Total Knee Arthroplasty: A Prospective Randomized Trial
Brief Title: Topical Anesthesia for Removal of Stitches After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201505116MINA
Record Dates: First submitted 2016-04-17; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Metal Staple Removal After Total Knee Replacement
Keywords: Total Knee Replacement; Stitch; Removal; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine patch (Experimental): The patients was randomly assigned to experimental group or placebo group. In this arm, lidocaine patches will be applied to the skin surrounding the surgical wound by one nurse practitioner. After more than 20 minutes the patch will be removed. Another nurse practitioner (double blinded) will remove the metal staples and record pain scale.
  Interventions: Drug: Lidocaine patch
- Placebo (Placebo Comparator): The patients was randomly assigned to experimental group or placebo group. In this arm, a placebo patch will be applied to the skin surrounding the surgical wound by one nurse practitioner. After more than 20 minutes the patch will be removed. Another nurse practitioner (double blinded) will remove the metal staples and record pain scale.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lidocaine patch — Lidocain patch will be applied around the surgical wound about 20 minutes before removal of staples.
  Arms: Lidocaine patch
Drug: placebo — Placebo patch will be applied around the surgical wound about 20 minutes before removal of staples.
  Arms: Placebo

SUMMARY:
Lidocaine patch is a safe and effective topical anesthetic agent for removal of metal staples after total knee replacement

DETAILED DESCRIPTION:
This is a double-blind randomised control trial. After informed consent, the patients who undergoes primary total knee replacement will be assigned to either control group or experimental group randomly. The effectiveness and complication will be analysed.

If the patients are not medically fit for the study (including contraindications for lidocaine), they will be excluded.

ELIGIBILITY:
Inclusion criteria:

1. Males and females, aged 50-100 years
2. The patients who undergo primary total knee replacement (performed by the same surgeon, Dr.Jiang)
3. Clear consciousness
4. No contraindication for staple removal on the post-operative day 7

Exclusion criteria:

1. Allergy to lidocaine
2. Patient with second or third degree atrio-ventricular block
3. Patients with severe Sinoatrial node block
4. Patients taking class I antiarrhythmia drugs
5. Pregnant patients
6. Patients undergoing revision total knee replacement
7. Contraindication for removal of staples on post-operative day 7

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale for pain | 30min
  The person who removes the staples evaluated the pain intensity. The pain intensity is evaluated with visual analog scale for pain

SECONDARY OUTCOMES:
Complication rate of lidocaine patch | Two weeks
  The incidence of related complications after application of lidocaine patch

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Chuan Jiang, Principal Investigator — Department of Orthopedic Surgery, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided